CLINICAL TRIAL: NCT04816188
Title: Heel Pain in Adolescents: A Pilot Study on the Effectiveness of Exercise Therapy and Activity Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Karin Silbernagel, Professor, University of Delaware
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1652996
Record Dates: First submitted 2021-03-18; First posted 2021-03-25 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Sever's Disease; Achilles Tendinopathy; Insertional Achilles Tendinopathy; Apophysitis; Calcaneus
Keywords: Achilles tendon; Pain; Activity modification; Sever's disease; Achilles tendinopathy; Apophysitis; Exercise
MeSH Terms: conditions — Pain; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise and Activity Modification (Experimental)
  Interventions: Other: Exercise Therapy and Activity Modification

INTERVENTIONS:
Other: Exercise Therapy and Activity Modification — Daily lower leg strengthening exercises Therapy and pain-guided activity modification.

SUMMARY:
Invesigators plan to conduct a 12-week longitudinal cohort study of 30 subjects with calcaneal apophysitis. Subjects will be included if they are between 7-17 years-old, have experienced an insidious onset of heel pain with running or jumping activities, and have no underlying diagnosis predisposing heel pain and no other injury that limits their ability to run and jump. Parents of subjects will be invited to participate by completing questionnaires related to their perspective of their child's symptoms, physical activity level, quality of life, and their satisfaction with the treatment protocol. Subjects will be asked to attend 4 monthly sessions consisting of evaluation and treatment.

DETAILED DESCRIPTION:
Investigators will recruit 30 subjects between ages 7-17 with heel pain and also invite their parent/guardian to participate in this research study. Participants will be evaluated at baseline, 4-weeks, 8-weeks and 12-weeks. Data collections at each assessment visit will be identical except for the baseline visit. The baseline evaluation will consist of questionnaires related to past medical history in addition to all other procedures. All evaluations will include patient-reported outcome measures, clinical measures, and measurement of tendon structure, mechanical properties, and muscle-tendon function Treatment sessions will occur immediately following the evaluation sessions (4 total). During treatment sessions, participants will be provided with education, therapeutic exercise instruction, and discussion of their training diary and home exercise program. Treatment sessions will last 30-45 minutes. In addition to the 4 in-person treatment sessions, virtual visits will take place 2 weeks in between each in-person visits, (one virtual visit maximum every 4 weeks) as needed. Virtual visits will be no longer than 30 minutes to discuss patient needs.

ELIGIBILITY:
Inclusion Criteria:

* Insidious onset of heel pain with running or jumping activities lasting at least three weeks
* Location of pain is focal at the calcaneus over the Achilles tendon attachment and/or the Achilles tendon

Exclusion Criteria:

* Subjects having an underlying diagnosis predisposing to heel pain (spina bifida, osteogenesis imperfecta, Larsen syndrome, cerebral palsy)
* History of calcaneal fracture or foot/ankle surgery in the past 6 months
* Another injury that limits the ability to perform exercises on the injured leg

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment - Achilles (VISA-A) questionnaire | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 6-weeks, 8-weeks,10-weeks and 12-weeks
  The VISA-A was specifically designed to assess symptom severity in individuals with Achilles tendinopathy and has demonstrated validity, reliability and responsiveness. Scores range from 0-100, where a higher score indicates less pain and symptoms with activity. This outcome measure has been used in previous trials with adolescents.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Pain Interference Scale | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 6-weeks, 8-weeks,10-weeks and 12-weeks
  The PROMIS Pain Interference Scale assesses symptom severity and pain with daily activity. Raw scores range from 8-40, where lower scores indicate less pain interference.
Tendon Structure | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 8-weeks, and 12-weeks
  Ultrasound images will be obtained using the LOGIQ e Ultrasound (GE Healthcare) system using a wide-band linear array probe (5.0-13.0 MHz). The subject will be prone lying with the hips and knees straight and the ankles hanging outside the treatment table. Three longitudinal images where the calcaneal insertion and as much of the tendon is visible will be saved. Three extended field of view images of the tendon between the insertion to the calcaneus and the start of the soleus muscle will be saved. Longitudinal and cross-sectional images will be taken at the area of tenderness to palpation on the injured side and at the same position on the contralateral side. These images will be used to evaluate tendon thickening, cross-sectional area, and the occurrence of hypoechoic areas.
Tendon Mechanical Properties | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 8-weeks, and 12-weeks
  Subjects will be examined using continuous shear wave elastography (cSWE). This is a non-invasive technique that uses a low-amplitude vibration to mechanically perturbate the tendon. The resultant shear wave is imaged using ultrasound. The area of maximum tendon pathology will be identified using palpation and B mode ultrasound imaging. The distance from calcaneal insertion to this area will be measured to allow for identification of a comparable location on the asymptomatic side as well as to ensure the same area is assessed at each follow-up. The ultrasound probe for cSWE will be placed at this location and the actuator will be placed just proximal to the ultrasound probe.
Muscle-Tendon Function | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 8-weeks, and 12-weeks
  Muscle-tendon function will be assessed by a functional test battery including a single-leg counter movement jump (CMJ), a single-leg drop CMJ, single-leg hopping, and the heel-rise endurance test. For jump tests, the jump height for three trials will be recorded using a light mat (MuscleLab®, Ergotest Innovations, Porsgrunn, Norway). The drop CMJ jump is performed on single leg by jumping from a 20cm high box, landing, and immediately jumping up for maximum height. Hopping is similar or jumping rope on one foot; two trials of 20 hops will be recorded using a light mat to calculate hop frequency, average height, and plyometric quotient (flight time / contact time). The heel-rise endurance test is a single-leg standing heel-rise test. The heel-rise test for endurance is performed on one leg at a time with the participant standing on a box with an incline of 10°. A metronome is used to maintain the frequency of 30 heel-rises per minute.
Compliance | Average compliance rate for each group over first year of study recruitment
  Compliance will be tracked using training diaries. The number of training diaries and prescribed exercise sessions completed, and days in adherence with activity modification guidelines will be recorded. Compliance rates will be reported as a percentage, relative to the participants duration of participation in the study.

SECONDARY OUTCOMES:
PROMIS Pediatric Global Health questionnaire | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 6-weeks, 8-weeks,10-weeks and 12-weeks
  The PROMIS Pediatric Global Health questionnaire will be used to assess self-reported impact of injury on mental and physical health. Raw scores range from 7-35, where higher scores indicate higher physical and mental health.
PROMIS Pediatric Physical Activity Short Form questionnaire | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 6-weeks, 8-weeks,10-weeks and 12-weeks
  The PROMIS Pediatric Physical Activity Short Form questionnaire will be used to assess self-reported capability over a 7 day period. Raw scores range from 8-40, where a higher score indicates higher physical activity levels.
The Foot and Ankle Outcomes Score (FAOS) | Change over time with evaluations at baseline, 2-weeks, 4-weels, 6-weeks, 8-weeks,10-weeks and 12-weeks
  Three subscales from The Foot and Ankle Outcomes Score (FAOS) will be used to measure foot and ankle-related quality of life (FOAS-QoL), symptoms (FAOS-S), and function in sport and recreation. Each subscale ranges from 0-100, where higher scores indicate better outcomes.
The Fear of Pain Questionnaire Child Report (FOBQC) | Change over time with evaluations at baseline, 2-weeks, 4-weels, 6-weeks, 8-weeks,10-weeks and 12-weeks
  The Fear of Pain Questionnaire Child Report (FOBQC) will assess fear of pain and avoidance of activities. Scores range from 0-96, where 0-34 indicates low fear and 51-96 indicates high fear.
The Global Rating of Change (GROC) scale | Change over time with evaluations at baseline, 2-weeks, 4-weels, 6-weeks, 8-weeks,10-weeks and 12-weeks
  The Global Rating of Change (GROC) scale, will be used to measure their satisfaction and perceived recovery of their child using a 10-point likert respectively ranging from -5 to +5 indicating a range between "not satisfied" to "very satisfied" and "much worse" to "much improved".
PROMIS Parent Proxy Pain Intensity questionnaire | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 6-weeks, 8-weeks,10-weeks and 12-weeks
  PROMIS Parent Proxy Pain Intensity will assess symptom severity from the parent's perspective. Parents are asked to rate their child's pain at it's worst on a scale of 0-10, where 0 is "no pain" and 10 is "worst pain imaginable".
PROMIS Parent Proxy Pain Interference questionnaire | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 6-weeks, 8-weeks,10-weeks and 12-weeks
  The PROMIS Parent Proxy Pain Interference Scale assesses symptom severity and pain with daily activity from the parent's perspective. Raw scores range from 8-40, where lower scores indicate less pain interference.
PROMIS Parent Proxy Global Health questionnaire | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 6-weeks, 8-weeks,10-weeks and 12-weeks
  The PROMIS Parent Proxy Global Health questionnaire will assess the parent's perspective on the participant's mental and physical health. Raw scores range from 7-35, where higher scores indicate higher physical and mental health.
PROMIS Parent Proxy Physical Activity questionnaire | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 6-weeks, 8-weeks,10-weeks and 12-weeks
  The PROMIS Parent Proxy Physical Activity form will be used to assess parent-reported capability of their child's physical activities over a 7 day period. Raw scores range from 4-20, where a higher score indicates higher physical activity level.
Fear of Pain Questionnaire Parent Report (FOBQP) | Change over time with evaluations at baseline, 2-weeks, 4-weeks, 6-weeks, 8-weeks,10-weeks and 12-weeks
  The Fear of Pain Questionnaire Parent Report (FOBQP) is a parent inventory to assess child pain-related fears. Scores range from 0-96, where 0-34 indicates low fear and 51-96 indicates high fear.
Ankle range of motion | Change over time with evaluations at baseline, 4-weeks, 8-weeks,10-weeks, and 12-weeks
  Ankle range of motion in non-weight bearing and weight bearing positions will be measured with a goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- STAR Building, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rachel JN, Williams JB, Sawyer JR, Warner WC, Kelly DM. Is radiographic evaluation necessary in children with a clinical diagnosis of calcaneal apophysitis (sever disease)? J Pediatr Orthop. 2011 Jul-Aug;31(5):548-50. doi: 10.1097/BPO.0b013e318219905c. PMID 21654464
- [Background] Robinson JM, Cook JL, Purdam C, Visentini PJ, Ross J, Maffulli N, Taunton JE, Khan KM; Victorian Institute Of Sport Tendon Study Group. The VISA-A questionnaire: a valid and reliable index of the clinical severity of Achilles tendinopathy. Br J Sports Med. 2001 Oct;35(5):335-41. doi: 10.1136/bjsm.35.5.335. PMID 11579069
- [Background] Suryavanshi JR, Goto R, Jivanelli B; PRiSM Outcomes Measures Research Interest Group; Aberdeen J, Duer T, Lam KC, Franklin CC, MacDonald J, Shea KG, Fabricant PD. Age-Appropriate Pediatric Sports Patient-Reported Outcome Measures and Their Psychometric Properties: A Systematic Review. Am J Sports Med. 2019 Nov;47(13):3270-3276. doi: 10.1177/0363546518818822. Epub 2019 Jan 16. PMID 30649907
- [Background] Rathleff MS, Graven-Nielsen T, Holmich P, Winiarski L, Krommes K, Holden S, Thorborg K. Activity Modification and Load Management of Adolescents With Patellofemoral Pain: A Prospective Intervention Study Including 151 Adolescents. Am J Sports Med. 2019 Jun;47(7):1629-1637. doi: 10.1177/0363546519843915. Epub 2019 May 16. PMID 31095417
- [Background] Forrest CB, Bevans KB, Pratiwadi R, Moon J, Teneralli RE, Minton JM, Tucker CA. Development of the PROMIS (R) pediatric global health (PGH-7) measure. Qual Life Res. 2014 May;23(4):1221-31. doi: 10.1007/s11136-013-0581-8. Epub 2013 Nov 22. PMID 24264804
- [Background] Roos EM, Brandsson S, Karlsson J. Validation of the foot and ankle outcome score for ankle ligament reconstruction. Foot Ankle Int. 2001 Oct;22(10):788-94. doi: 10.1177/107110070102201004. PMID 11642530
- [Background] Simons LE, Sieberg CB, Carpino E, Logan D, Berde C. The Fear of Pain Questionnaire (FOPQ): assessment of pain-related fear among children and adolescents with chronic pain. J Pain. 2011 Jun;12(6):677-86. doi: 10.1016/j.jpain.2010.12.008. Epub 2011 Feb 26. PMID 21354866
- [Background] Silbernagel KG, Shelley K, Powell S, Varrecchia S. Extended field of view ultrasound imaging to evaluate Achilles tendon length and thickness: a reliability and validity study. Muscles Ligaments Tendons J. 2016 May 19;6(1):104-10. doi: 10.11138/mltj/2016.6.1.104. eCollection 2016 Jan-Mar. PMID 27331037
- [Background] Zellers JA, Bley BC, Pohlig RT, Alghamdi NH, Silbernagel KG. FREQUENCY OF PATHOLOGY ON DIAGNOSTIC ULTRASOUND AND RELATIONSHIP TO PATIENT DEMOGRAPHICS IN INDIVIDUALS WITH INSERTIONAL ACHILLES TENDINOPATHY. Int J Sports Phys Ther. 2019 Sep;14(5):761-769. PMID 31598414
- [Background] Cortes DH, Suydam SM, Silbernagel KG, Buchanan TS, Elliott DM. Continuous Shear Wave Elastography: A New Method to Measure Viscoelastic Properties of Tendons in Vivo. Ultrasound Med Biol. 2015 Jun;41(6):1518-29. doi: 10.1016/j.ultrasmedbio.2015.02.001. Epub 2015 Mar 19. PMID 25796414
- [Background] Silbernagel KG, Gustavsson A, Thomee R, Karlsson J. Evaluation of lower leg function in patients with Achilles tendinopathy. Knee Surg Sports Traumatol Arthrosc. 2006 Nov;14(11):1207-17. doi: 10.1007/s00167-006-0150-6. Epub 2006 Jul 21. PMID 16858560
- [Background] Silbernagel KG, Thomee R, Eriksson BI, Karlsson J. Continued sports activity, using a pain-monitoring model, during rehabilitation in patients with Achilles tendinopathy: a randomized controlled study. Am J Sports Med. 2007 Jun;35(6):897-906. doi: 10.1177/0363546506298279. Epub 2007 Feb 16. PMID 17307888